CLINICAL TRIAL: NCT05588479
Title: Effects of Pomegranate Extract on Inflammatory Markers, Physical and Cognitive Function and Cardiometabolic Risk Factors in Older Adults: a Randomised Parallel Trial
Brief Title: Pomegranate Extract and Inflammageing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester Metropolitan University (Other)
Responsible Party: Principal Investigator, Grace Farhat, Senior lecturer in Nutrition and Dietetics, Manchester Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 47627
Record Dates: First submitted 2022-10-12; First posted 2022-10-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Aging
MeSH Terms: interventions — pomegranate fruit rind

STUDY DESIGN:
Intervention Model Description: Two-arm double blind parallel trial where participants will be randomly assigned to receive either placebo capsules (control) or pomegranate extract capsules (740 mg) for 12 weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: Capsules were masked by the manufacturer and blinded to outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Capsules with no pomegranate extract One capsule to be administered once a day for 12 weeks.
  Interventions: Dietary Supplement: Control
- Intervention (Experimental): Capsules with 740 mg of pomegranate extract Two capsules to be administered once a day for 12 weeks.
  Interventions: Dietary Supplement: Pomegranate extract

INTERVENTIONS:
Dietary Supplement: Pomegranate extract — Two capsules of pomegranate extract (740 mg) will be taken daily at any time of the day for a period of 12 weeks.
  Arms: Intervention
Dietary Supplement: Control — One capsule of containing no pomegranate extract will be taken daily at any time of the day for a period of 12 weeks.
  Arms: Control

SUMMARY:
The growing ageing population has resulted in an increase in the prevalence of frailty, cognitive disorders and cardiovascular diseases, representing a major cause of disability in older adults. Inflammation has been suggested as a pivotal factor leading to these disorders and is exacerbated by obesity. Polyphenols are antioxidants and anti-inflammatory agents that have been previously linked to a decrease in inflammation and cardiometabolic risk factors and an improvement in physical and cognitive function, yet research remain limited and inconclusive. This study aims to assess the effect of daily pomegranate extract supplementation on inflammatory response, cognitive and physical function and cardiometabolic risk factors in older adults. Seventy-one normal weight and overweight participants (55-70 years) will be assigned to consume either pomegranate extract capsules or placebo capsules for 12 weeks. Anthropometric measures (weight, height, waist circumference and hip circumference), body composition, blood pressure and a fasted venous blood sample will be collected during each visit at baseline, week 6 & week 12. Participants will also undergo computerised cognitive tests and physical function tests. Inflammatory markers, telomerase activity, serum glucose and lipid levels will be analysed. Diet diaries will be collected 3 times (at baseline, week 6 & week 12) during the intervention. This study will help elucidate the effects of pomegranate supplementation and inform future longitudinal trials looking at the combination of antioxidants and other lifestyle factors (such as physical activity) on the promotion of well-being and healthy ageing.

DETAILED DESCRIPTION:
After signing an informed consent, participants will be asked to attend the Physiology Lab at Manchester Metropolitan University at baseline, week 6 and week 12. Anthropometric measures (weight, height, waist circumference and hip circumference) will be collected during each visit, and body composition will be measured using air displacement plethysmography (BOD POD®). Blood pressure will be measured 3 times after a 10-minute rest based on the World Health Organisation (WHO) protocol and a fasted venous blood sample (20 ml) will be collected. Participants will then undergo physical assessment tests (to assess standing balance, gait speed, and chair sit to stand) and computerised cognitive tests (to assess executive function, memory, vigilance and attention).

Participants will also answer a general demographic and lifestyle questionnaire during the first visit. To control for changes in the diet, they will be asked to fill a paper-based 3-day food diary 3 times (at baseline, week 6 & week 12) during the intervention. Food diaries will be analysed using Nutritics (v.4) dietary analysis software.

ELIGIBILITY:
Inclusion Criteria:

Age 55-70 years; Normal weight (BMI 18.5-24.9 Kg/m2) and overweight (BMI 25- 29.9 Kg/m2); All genders; No diagnosed metabolic diseases.

Exclusion Criteria:

Participants who have been on a weight loss regimen over the past 2 months, those with diagnosed chronic disease (diabetes, cardiovascular disease (CVD), renal disease etc…) or taking any medications that could modulate inflammation (statins etc..).

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 (IL-6) levels | Baseline, week 6 & week 12
  Changes in IL-6 levels will be measured in a fasted blood sample using a commercially available assay kit.

SECONDARY OUTCOMES:
CRP (C-reactive protein) levels | Baseline, week 6 & week 12
  Changes in CRP levels will be measured in a fasted blood sample using a commercially available assay kit.
Interleukin 1 (IL-1) levels | Baseline, week 6 & week 12
  Changes in IL-1 levels will be measured in a fasted blood sample using a commercially available assay kit.
Interleukin 2 (IL-2) levels | Baseline, week 6 & week 12
  Changes in IL-2 levels will be measured in a fasted blood sample using a commercially available assay kit.
Insulin growth factor-1 (IGF-1) levels | Baseline, week 6 & week 12
  Changes in IGF-1 levels will be measured in a fasted blood sample using a commercially available assay kit.
Tumour necrosis factor (TNF-α) levels | Baseline, week 6 & week 12
  Changes in TNF-α levels will be measured in a fasted blood sample using a commercially available assay kit.
Plasminogen Activator Inhibitor-1 (PAI-1) levels | Baseline, week 6 & week 12
  Changes in PAI-1 levels will be measured in a fasted blood sample using a commercially available assay kit.
Telomerase activity | Baseline, week 6 & week 12
  Changes in telomerase activity will be measured in a fasted blood sample using a commercially available assay kit.
Corsi block-tapping test | Baseline, week 6 & week 12
  Changes in working memory will be assessed using Corsi block-tapping computerised cognitive test.
Rey Verbal Learning test | Baseline, week 6 & week 12
  Changes in working memory will be assessed using Rey Verbal Learning computerised cognitive test.
Tower of Hanoi test | Baseline, week 6 & week 12
  Changes in executive function will be assessed using Tower of Hanoi computerised cognitive test.
Wisconsin test | Baseline, week 6 & week 12
  Changes in executive function will be assessed using Wisconsin computerised cognitive test.
Stroop test | Baseline, week 6 & week 12
  Changes in executive function will be assessed using Stroop computerised cognitive test.
Digits span test | Baseline, week 6 & week 12
  Changes in working memory will be assessed using Digits span computerised cognitive test.
Hand grip strength | Baseline, week 6 & week 12
  Changes in muscle strength will be assessed using hand grip strength physical test.
Standing balance | Baseline, week 6 & week 12
  Changes in muscle function will be assessed using standing balance physical test.
Gait speed | Baseline, week 6 & week 12
  Changes in muscle function will be assessed using gait speed physical test.
Chair sit to stand | Baseline, week 6 & week 12
  Changes in muscle function will be assessed using chair sit to stand physical test.
Fasting serum glucose levels | Baseline, week 6 & week 12
  Changes in glucose levels will be measured in a fasted blood sample using a commercially available assay kit.
Fasting lipid levels | Baseline, week 6 & week 12
  Changes in lipid levels (TC, HDL, LDL & TG) will be measured in a fasted blood sample using a commercially available assay kit.
Blood pressure | Baseline, week 6 & week 12
  Changes in blood pressure will be Blood pressure will be measured 3 times after a 10-minute rest based on the WHO protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Metropolitan University school of Health sciences, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No